CLINICAL TRIAL: NCT03977870
Title: Identification of New Genetic Markers for the Risk of Recurrence of Venous Thromboembolism by Whole Genome Analysis: Case-control Study Nested in the MARTHA Cohort
Brief Title: Identification of New Genetic Markers for the Risk of Recurrence of Venous Thromboembolism by Whole Genome Analysis
Acronym: MARTHARecidive
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-27
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Venous Thromboembolism (VTE)
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Venous thromboembolism (VTE)
  Interventions: Other: vital status determination

INTERVENTIONS:
Other: vital status determination — consultation of national registries

SUMMARY:
Venous thromboembolism (VTE) is a common and potentially fatal pathology in France. The risk of recurrence is around 5 to 7% per year. The identification of patients at risk of VTE and its prevention is a real health issue in particular. 50% of MTEV recurrences occur in the absence of a risk situation, suggesting the involvement of specific risk factors for MTEV recurrence that have not been identified to date.

In the last ten years, so-called "genome-whole" or "genome wide" association (GWAS) approaches have identified new genetic risk factors for the first episode of VTE. On the other hand, no study has focused on the predictive factors of recurrence.

The previous project, conducted from 2012 (NCT02904967), had as its main objective to identify new genes for susceptibility to MTEV recurrence by comparing cases of MTEV recurrence versus controls having had a single episode of MTEV. The MARTHA cohort (1,542 patients) is extremely valuable study material and is one of the few cohorts in the world with genome-wide data in the field of VTE. Follow-up could only be performed in 359 patients, 76 (21%) of whom presented with a new episode of VTE.

The objective of this project is to increase the number of patients for whom the investigators will have information on recurrence / non-recurrence of VTE, by querying national registries on the vital status of patients, and possible causes of death. .

These new data on the occurrence or not of a new thrombotic episode, will be confronted with the genetic data already available in all the patients in order to identify specific genetic risk factors and potentially predictive of the recurrence of MTEV.

ELIGIBILITY:
Inclusion Criteria:

* patients of the MARTHA cohort

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Martha cohort is composed of 1542 subjects from the Region of Marseille with at least one episode of VTE documented. Patients in the MARTHA cohort have already all been genotyped for approximately 500,000 polymorphisms
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
MTEV recurrence | 12 months
  information on recurrence / non-recurrence of VTE, by querying national registries on the vital status of patients, and possible causes of death.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido Pradalié, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France